CLINICAL TRIAL: NCT03750747
Title: Assessing the Feasibility and Effectiveness of Introducing Pulse Oximetry in IMCI Services to Manage Acute Respiratory Infections at First Level Health Facilities of Bangladesh
Brief Title: Assessing the Feasibility and Effectiveness of Introducing Pulse Oximetry in IMCI Services
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-18054
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Childhood Pneumonia; Hypoxemia
Keywords: IMCI services; Pulse Oximeter; Acute respiratory infections; Implementation research; Hypoxaemia; Childhood Pneumonia; Resource poor settings
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Pulse Oximeter) (Experimental): The intervention facilities will provide IMCI services with PO in addition to following existing IMCI guidelines. The IMCI service providers will classify and treat children presenting with cough and difficult breathing based on history and clinical signs. In addition, they will use PO to measure the SpO2 status of the sick children. Children clinically classified as 'Pneumonia' but having SpO2<90% will be referred to higher-level facilities for in-patient management. Only the children clinically classified 'Pneumonia' and having SpO2>90% will be treated through home-based management with oral antibiotics (amoxicillin, twice daily for five day).
  Interventions: Device: Pulse Oximeter
- Comparison (No Intervention): The comparison facilities will continue providing routine IMCI services as per the existing guidelines. In routine IMCI services, IMCI service providers classify and treat children presenting with cough and difficult breathing based on history and clinical signs only. In routine IMCI services in Bangladesh, PO has not been introduced. Therefore, in the comparison facilities all children clinically classified as 'Pneumonia' will be treated through home-based management with oral antibiotics (amoxicillin, twice daily for five day)

INTERVENTIONS:
Device: Pulse Oximeter — SpO2 will be measured using a handheld PO device (selected for this study) applying the low noise cabled sensor. For patients weighing <10 kg, the sensor will be placed on the big toe. For patients weighing >10 kg, the sensor will be placed on an index finger. In case of failure in the first attempt, the alternate toe or index finger will be tried (second attempt). First, the sensor will be placed on toe or index finger and then the PO will be powered-on. A stable Sp02 reading will be considered to be obtained if SpO2 reading is stable by ±1 % for at least 10 seconds and the device signal strength is displayed to be adequate (green signal). Second attempt will be warranted if a stable reading is not obtaining within 1-2 minutes.
  Arms: Intervention (Pulse Oximeter)

SUMMARY:
The purpose of the study is to assess the feasibility, acceptability and operational challenges of introducing Pulse Oximeter (PO) in IMCI services to manage acute respiratory infections at first-level primary care facilities in Bangladesh (phase 1). The investigators will also evaluate the effectiveness and cost-effectiveness of introducing PO in IMCI services at first level primary care health facilities (phase 2).

This study will employ a cluster randomized controlled trial design to evaluate the effectiveness of introducing PO in IMCI services (phase-2 objective). The feasibility assessment (phase-1 objective) will be nested within the larger effectiveness trail as internal piloting; which will help in generating evidence for designing a robust phase-2 trial. First-level primary healthcare facilities providing IMCI services will be regarded as clusters and the unit of randomization. Sixteen first level primary care health facilities (UH&FWC) will be randomly assigned to comparison and intervention facilities.

DETAILED DESCRIPTION:
Background:

1. Burden: Pneumonia is the leading cause of childhood mortality which accounts for 16% of all under-5 deaths in Bangladesh and globally. Most of these deaths happen in the developing countries, where WHO recommends adopting Integrated Management of Childhood Illness (IMCI) as a strategy for outpatient management of common childhood illnesses, including pneumonia, in these poor resource settings.
2. Knowledge gap: As per the IMCI guidelines, 'Pneumonia' can be treated through home-based management with oral antibiotics, whereas 'Severe Pneumonia' should be referred to high-level facilities for inpatient care. Previously, chest indrawing was considered as one of the signs of 'Severe Pneumonia.' In 2014, WHO revised the IMCI guidelines recommending chest indrawing as a sign of 'Pneumonia' instead of 'Severe Pneumonia.' A systematic review of the home-based management of chest indrawing 'Pneumonia' reported a treatment failure rate of 8.5% on day 6. This implies that some of the chest indrawing 'Pneumonia' cases will require special inpatient care in addition to oral antibiotics and home-based management as currently recommended by WHO.
3. Relevance: Hypoxemia (SpO2<90%) is one of the strongest predictors of mortality due to pneumonia. Many of the chest indrawing 'Pneumonia' cases may have hypoxemia and need specialized inpatient care. In response to this, WHO recommended measuring SpO2 level with pulse oximetry (PO) as a part of IMCI services. As per the updated IMCI guidelines, any sick child (2-59 months) having SpO2 <90% should be referred for inpatient management, irrespective of its clinical classification. However, most of the primary care facilities are devoid of PO; and there is a paucity of evidence related to the feasibility and effectiveness of introducing of PO in primary care facilities.

Objectives:

* Phase-1: To assess the feasibility, acceptability and operational challenges of introducing PO in IMCI services at first-level primary care health facilities in Bangladesh
* Phase-2: To evaluate the effectiveness and cost-effectiveness of introducing PO in IMCI services at first level primary care health facilities in Bangladesh

Methods:

This study will employ a cluster randomized controlled trial design to evaluate the effectiveness of introducing PO in IMCI services (phase-2 objective). The feasibility assessment (phase-1 objective) will be nested within the larger effectiveness trail as an internal piloting; which will help in generating evidence for designing a robust phase-2 trial. First-level primary healthcare facilities providing IMCI services will be regarded as clusters and the unit of randomization. Twenty-four first level primary care health facilities will be randomly assigned to comparison and intervention facilities.

In phase-1, the feasibility, acceptability and operational challenges of introducing PO in IMCI services will be assessed in the intervention facilities. Structured observation of the use of PO in IMCI services and community case tracking will be conducted to address the phase-1 objective. Rigorous process documentation and qualitative method of data collection will be employed to document the process of implementation and assess implementation outcomes.

In phase-2, effectiveness will be assessed through community case tracking in both comparison and intervention facilities. Treatment failure rate will be the primary outcome and the analysis will consider 'intention to treat' approach. In addition, activity-based costing method will be adopted for collecting cost-related data.

Outcome measures/variables:

This study will assess the effectiveness of integrating PO in IMCI services in first-level health facilities in Bangladesh. PO will be able to identify children who are classified as 'Pneumonia' based on history and clinical signs but have hypoxaemia. It will facilitate referral of children with hypoxaemia to higher level facilities.

ELIGIBILITY:
Inclusion Criteria:

1. Sick children aged 2 to 59 months
2. Presenting with cough or difficult breathing
3. Receiving IMCI services in the selected facilities will be enrolled

Exclusion Criteria:

1. Severely ill children who need to be referred immediately
2. If the parents of the children are unwilling to participate

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 612 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate | up to 12 months
  The primary outcome of interest is treatment failure rate among those who are clinically classified as 'Pneumonia'. Operational definition of treatment failure will be finalized based on expert consultation and opinion of the caretakers of sick children through PPI. For illustrative purpose, an operational definition of the treatment failure is presented below which is based on some similar studies, i.e. SAT, AFRINEST, NO-SHOT, etc.Presence of any of the followings signs on day-6 and day-12 will be a considered as treatment failure:
  * Death
  * Appearance of any of the danger signs:
    * Inability to drink
    * Vomits everything
    * Lethargy or unconsciousness
    * Convulsions or history of convulsion
  * Persistence of
    * Low oxygen saturation (SpO2<90%)
    * Chest indrawing
    * Fast breathing

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ehsanur Rahman, MBBS, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Confidentiality of the data will be ensured at all steps of the study including data collection, data management, access to data and use of the information. All personal identifiers will be removed from the data prior to analysis.

REFERENCES:
- [Background] Liu L, Oza S, Hogan D, Chu Y, Perin J, Zhu J, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of under-5 mortality in 2000-15: an updated systematic analysis with implications for the Sustainable Development Goals. Lancet. 2016 Dec 17;388(10063):3027-3035. doi: 10.1016/S0140-6736(16)31593-8. Epub 2016 Nov 11. PMID 27839855
- [Background] Lim YW, Steinhoff M, Girosi F, Holtzman D, Campbell H, Boer R, Black R, Mulholland K. Reducing the global burden of acute lower respiratory infections in children: the contribution of new diagnostics. Nature. 2006 Nov 23;444 Suppl 1:9-18. doi: 10.1038/nature05442. No abstract available. PMID 17159890
- [Background] Sazawal S, Black RE; Pneumonia Case Management Trials Group. Effect of pneumonia case management on mortality in neonates, infants, and preschool children: a meta-analysis of community-based trials. Lancet Infect Dis. 2003 Sep;3(9):547-56. doi: 10.1016/s1473-3099(03)00737-0. PMID 12954560
- [Background] Arifeen SE, Hoque DM, Akter T, Rahman M, Hoque ME, Begum K, Chowdhury EK, Khan R, Blum LS, Ahmed S, Hossain MA, Siddik A, Begum N, Sadeq-ur Rahman Q, Haque TM, Billah SM, Islam M, Rumi RA, Law E, Al-Helal ZA, Baqui AH, Schellenberg J, Adam T, Moulton LH, Habicht JP, Scherpbier RW, Victora CG, Bryce J, Black RE. Effect of the Integrated Management of Childhood Illness strategy on childhood mortality and nutrition in a rural area in Bangladesh: a cluster randomised trial. Lancet. 2009 Aug 1;374(9687):393-403. doi: 10.1016/S0140-6736(09)60828-X. PMID 19647607
- [Background] Chowdhury EK, El Arifeen S, Rahman M, Hoque DE, Hossain MA, Begum K, Siddik A, Begum N, Sadeq-ur Rahman Q, Akter T, Haque TM, Al-Helal ZM, Baqui AH, Bryce J, Black RE. Care at first-level facilities for children with severe pneumonia in Bangladesh: a cohort study. Lancet. 2008 Sep 6;372(9641):822-30. doi: 10.1016/S0140-6736(08)61166-6. Epub 2008 Aug 18. PMID 18715634
- [Background] Armstrong Schellenberg JR, Adam T, Mshinda H, Masanja H, Kabadi G, Mukasa O, John T, Charles S, Nathan R, Wilczynska K, Mgalula L, Mbuya C, Mswia R, Manzi F, de Savigny D, Schellenberg D, Victora C. Effectiveness and cost of facility-based Integrated Management of Childhood Illness (IMCI) in Tanzania. Lancet. 2004 Oct 30-Nov 5;364(9445):1583-94. doi: 10.1016/S0140-6736(04)17311-X. PMID 15519628
- [Background] Owais A, Sultana S, Stein AD, Bashir NH, Awaldad R, Zaidi AK. Why do families of sick newborns accept hospital care? A community-based cohort study in Karachi, Pakistan. J Perinatol. 2011 Sep;31(9):586-92. doi: 10.1038/jp.2010.191. Epub 2011 Jan 27. PMID 21273989
- [Background] Peterson S, Nsungwa-Sabiiti J, Were W, Nsabagasani X, Magumba G, Nambooze J, Mukasa G. Coping with paediatric referral--Ugandan parents' experience. Lancet. 2004 Jun 12;363(9425):1955-6. doi: 10.1016/S0140-6736(04)16411-8. PMID 15194257
- [Background] Addo-Yobo E, Chisaka N, Hassan M, Hibberd P, Lozano JM, Jeena P, MacLeod WB, Maulen I, Patel A, Qazi S, Thea DM, Nguyen NT. Oral amoxicillin versus injectable penicillin for severe pneumonia in children aged 3 to 59 months: a randomised multicentre equivalency study. Lancet. 2004 Sep 25-Oct 1;364(9440):1141-8. doi: 10.1016/S0140-6736(04)17100-6. PMID 15451221
- [Background] Hazir T, Fox LM, Nisar YB, Fox MP, Ashraf YP, MacLeod WB, Ramzan A, Maqbool S, Masood T, Hussain W, Murtaza A, Khawar N, Tariq P, Asghar R, Simon JL, Thea DM, Qazi SA; New Outpatient Short-Course Home Oral Therapy for Severe Pneumonia Study Group. Ambulatory short-course high-dose oral amoxicillin for treatment of severe pneumonia in children: a randomised equivalency trial. Lancet. 2008 Jan 5;371(9606):49-56. doi: 10.1016/S0140-6736(08)60071-9. PMID 18177775
- [Background] Straus WL, Qazi SA, Kundi Z, Nomani NK, Schwartz B. Antimicrobial resistance and clinical effectiveness of co-trimoxazole versus amoxycillin for pneumonia among children in Pakistan: randomised controlled trial. Pakistan Co-trimoxazole Study Group. Lancet. 1998 Jul 25;352(9124):270-4. doi: 10.1016/s0140-6736(97)10294-x. PMID 9690406
- [Background] Addo-Yobo E, Anh DD, El-Sayed HF, Fox LM, Fox MP, MacLeod W, Saha S, Tuan TA, Thea DM, Qazi S; Multicenter Amoxicillin Severe pneumonia Study (MASS) Group. Outpatient treatment of children with severe pneumonia with oral amoxicillin in four countries: the MASS study. Trop Med Int Health. 2011 Aug;16(8):995-1006. doi: 10.1111/j.1365-3156.2011.02787.x. Epub 2011 May 4. PMID 21545381
- [Background] Atkinson M, Lakhanpaul M, Smyth A, Vyas H, Weston V, Sithole J, Owen V, Halliday K, Sammons H, Crane J, Guntupalli N, Walton L, Ninan T, Morjaria A, Stephenson T. Comparison of oral amoxicillin and intravenous benzyl penicillin for community acquired pneumonia in children (PIVOT trial): a multicentre pragmatic randomised controlled equivalence trial. Thorax. 2007 Dec;62(12):1102-6. doi: 10.1136/thx.2006.074906. Epub 2007 Jun 13. PMID 17567657
- [Background] Ayieko P, English M. Case management of childhood pneumonia in developing countries. Pediatr Infect Dis J. 2007 May;26(5):432-40. doi: 10.1097/01.inf.0000260107.79355.7d. PMID 17468655
- [Background] Bari A, Sadruddin S, Khan A, Khan Iu, Khan A, Lehri IA, Macleod WB, Fox MP, Thea DM, Qazi SA. Community case management of severe pneumonia with oral amoxicillin in children aged 2-59 months in Haripur district, Pakistan: a cluster randomised trial. Lancet. 2011 Nov 19;378(9805):1796-803. doi: 10.1016/S0140-6736(11)61140-9. Epub 2011 Nov 10. PMID 22078721
- [Background] Fox MP, Thea DM, Sadruddin S, Bari A, Bonawitz R, Hazir T, Bin Nisar Y, Qazi SA; Pneumonia Studies Group. Low rates of treatment failure in children aged 2-59 months treated for severe pneumonia: a multisite pooled analysis. Clin Infect Dis. 2013 Apr;56(7):978-87. doi: 10.1093/cid/cis1201. Epub 2012 Dec 21. PMID 23264361
- [Background] Ahmed HM, Mitchell M, Hedt B. National implementation of Integrated Management of Childhood Illness (IMCI): policy constraints and strategies. Health Policy. 2010 Jul;96(2):128-33. doi: 10.1016/j.healthpol.2010.01.013. Epub 2010 Feb 21. PMID 20176407
- [Background] Walter ND, Lyimo T, Skarbinski J, Metta E, Kahigwa E, Flannery B, Dowell SF, Abdulla S, Kachur SP. Why first-level health workers fail to follow guidelines for managing severe disease in children in the Coast Region, the United Republic of Tanzania. Bull World Health Organ. 2009 Feb;87(2):99-107. doi: 10.2471/blt.08.050740. PMID 19274361
- [Background] Reed C, Madhi SA, Klugman KP, Kuwanda L, Ortiz JR, Finelli L, Fry AM. Development of the Respiratory Index of Severity in Children (RISC) score among young children with respiratory infections in South Africa. PLoS One. 2012;7(1):e27793. doi: 10.1371/journal.pone.0027793. Epub 2012 Jan 4. PMID 22238570
- [Background] Subhi R, Adamson M, Campbell H, Weber M, Smith K, Duke T; Hypoxaemia in Developing Countries Study Group. The prevalence of hypoxaemia among ill children in developing countries: a systematic review. Lancet Infect Dis. 2009 Apr;9(4):219-27. doi: 10.1016/S1473-3099(09)70071-4. PMID 19324294
- [Background] Nair H, Simoes EA, Rudan I, Gessner BD, Azziz-Baumgartner E, Zhang JSF, Feikin DR, Mackenzie GA, Moiisi JC, Roca A, Baggett HC, Zaman SM, Singleton RJ, Lucero MG, Chandran A, Gentile A, Cohen C, Krishnan A, Bhutta ZA, Arguedas A, Clara AW, Andrade AL, Ope M, Ruvinsky RO, Hortal M, McCracken JP, Madhi SA, Bruce N, Qazi SA, Morris SS, El Arifeen S, Weber MW, Scott JAG, Brooks WA, Breiman RF, Campbell H; Severe Acute Lower Respiratory Infections Working Group. Global and regional burden of hospital admissions for severe acute lower respiratory infections in young children in 2010: a systematic analysis. Lancet. 2013 Apr 20;381(9875):1380-1390. doi: 10.1016/S0140-6736(12)61901-1. Epub 2013 Jan 29. PMID 23369797
- [Background] Sherman B, Nisenboum JM, Jesberger BL, Morrow CA, Jesberger JA. Assessment of dysphagia with the use of pulse oximetry. Dysphagia. 1999 Summer;14(3):152-6. doi: 10.1007/PL00009597. PMID 10341112
- [Background] Schnapp LM, Cohen NH. Pulse oximetry. Uses and abuses. Chest. 1990 Nov;98(5):1244-50. doi: 10.1378/chest.98.5.1244. PMID 2225973
- [Background] Floyd J, Wu L, Hay Burgess D, Izadnegahdar R, Mukanga D, Ghani AC. Evaluating the impact of pulse oximetry on childhood pneumonia mortality in resource-poor settings. Nature. 2015 Dec 3;528(7580):S53-9. doi: 10.1038/nature16043. PMID 26633766
- [Background] Duke T, Subhi R, Peel D, Frey B. Pulse oximetry: technology to reduce child mortality in developing countries. Ann Trop Paediatr. 2009 Sep;29(3):165-75. doi: 10.1179/027249309X12467994190011. PMID 19689857
- [Background] Pedersen T, Dyrlund Pedersen B, Moller AM. Pulse oximetry for perioperative monitoring. Cochrane Database Syst Rev. 2003;(3):CD002013. doi: 10.1002/14651858.CD002013. PMID 12917918
- [Background] Schroeder AR, Marmor AK, Pantell RH, Newman TB. Impact of pulse oximetry and oxygen therapy on length of stay in bronchiolitis hospitalizations. Arch Pediatr Adolesc Med. 2004 Jun;158(6):527-30. doi: 10.1001/archpedi.158.6.527. PMID 15184214
- [Background] Dildy GA, van den Berg PP, Katz M, Clark SL, Jongsma HW, Nijhuis JG, Loucks CA. Intrapartum fetal pulse oximetry: fetal oxygen saturation trends during labor and relation to delivery outcome. Am J Obstet Gynecol. 1994 Sep;171(3):679-84. doi: 10.1016/0002-9378(94)90081-7. PMID 8092214
- [Background] Ramanathan R, Durand M, Larrazabal C. Pulse oximetry in very low birth weight infants with acute and chronic lung disease. Pediatrics. 1987 Apr;79(4):612-7. PMID 2434913
- [Background] Mallory MD, Shay DK, Garrett J, Bordley WC. Bronchiolitis management preferences and the influence of pulse oximetry and respiratory rate on the decision to admit. Pediatrics. 2003 Jan;111(1):e45-51. doi: 10.1542/peds.111.1.e45. PMID 12509594
- [Background] Mower WR, Sachs C, Nicklin EL, Safa P, Baraff LJ. Effect of routine emergency department triage pulse oximetry screening on medical management. Chest. 1995 Nov;108(5):1297-302. doi: 10.1378/chest.108.5.1297. PMID 7587433
- [Background] Reich JD, Miller S, Brogdon B, Casatelli J, Gompf TC, Huhta JC, Sullivan K. The use of pulse oximetry to detect congenital heart disease. J Pediatr. 2003 Mar;142(3):268-72. doi: 10.1067/mpd.2003.87. PMID 12640374
- [Background] Ewer AK, Middleton LJ, Furmston AT, Bhoyar A, Daniels JP, Thangaratinam S, Deeks JJ, Khan KS; PulseOx Study Group. Pulse oximetry screening for congenital heart defects in newborn infants (PulseOx): a test accuracy study. Lancet. 2011 Aug 27;378(9793):785-94. doi: 10.1016/S0140-6736(11)60753-8. Epub 2011 Aug 4. PMID 21820732
- [Background] Bierman MI, Stein KL, Snyder JV. Pulse oximetry in the postoperative care of cardiac surgical patients. A randomized controlled trail. Chest. 1992 Nov;102(5):1367-70. doi: 10.1378/chest.102.5.1367. PMID 1424853
- [Background] Abrams GA, Sanders MK, Fallon MB. Utility of pulse oximetry in the detection of arterial hypoxemia in liver transplant candidates. Liver Transpl. 2002 Apr;8(4):391-6. doi: 10.1053/jlts.2002.32252. PMID 11965585
- [Background] Brouillette RT, Morielli A, Leimanis A, Waters KA, Luciano R, Ducharme FM. Nocturnal pulse oximetry as an abbreviated testing modality for pediatric obstructive sleep apnea. Pediatrics. 2000 Feb;105(2):405-12. doi: 10.1542/peds.105.2.405. PMID 10654964
- [Background] Halevy A, Halpern Z, Negri M, Hod G, Weissgarten J, Averbukh Z, Modai D. Pulse oximetry in the evaluation of the painful hand after arteriovenous fistula creation. J Vasc Surg. 1991 Oct;14(4):537-9. PMID 1920651
- [Background] Tin W, Milligan DW, Pennefather P, Hey E. Pulse oximetry, severe retinopathy, and outcome at one year in babies of less than 28 weeks gestation. Arch Dis Child Fetal Neonatal Ed. 2001 Mar;84(2):F106-10. doi: 10.1136/fn.84.2.f106. PMID 11207226
- [Background] Anderson CG, Benitz WE, Madan A. Retinopathy of prematurity and pulse oximetry: a national survey of recent practices. J Perinatol. 2004 Mar;24(3):164-8. doi: 10.1038/sj.jp.7211067. PMID 14999216
- [Background] Rahman AE, Iqbal A, Hoque DM, Moinuddin M, Zaman SB, Rahman QS, Begum T, Chowdhury AI, Haider R, Arifeen SE, Kissoon N, Larson CP. Managing Neonatal and Early Childhood Syndromic Sepsis in Sub-District Hospitals in Resource Poor Settings: Improvement in Quality of Care through Introduction of a Package of Interventions in Rural Bangladesh. PLoS One. 2017 Jan 23;12(1):e0170267. doi: 10.1371/journal.pone.0170267. eCollection 2017. PMID 28114415
- [Background] Garde A, Zhou G, Raihana S, Dunsmuir D, Karlen W, Dekhordi P, Huda T, Arifeen SE, Larson C, Kissoon N, Dumont GA, Ansermino JM. Respiratory rate and pulse oximetry derived information as predictors of hospital admission in young children in Bangladesh: a prospective observational study. BMJ Open. 2016 Aug 17;6(8):e011094. doi: 10.1136/bmjopen-2016-011094. PMID 27534987
- [Background] Raihana S, Dunsmuir D, Huda T, Zhou G, Rahman QS, Garde A, Moinuddin M, Karlen W, Dumont GA, Kissoon N, El Arifeen S, Larson C, Ansermino JM. Correction: Development and Internal Validation of a Predictive Model Including Pulse Oximetry for Hospitalization of Under-Five Children in Bangladesh. PLoS One. 2016 Jan 15;11(1):e0147560. doi: 10.1371/journal.pone.0147560. eCollection 2016. No abstract available. PMID 26771879
- [Background] McCollum ED, King C, Deula R, Zadutsa B, Mankhambo L, Nambiar B, Makwenda C, Masache G, Lufesi N, Mwansambo C, Costello A, Colbourn T. Pulse oximetry for children with pneumonia treated as outpatients in rural Malawi. Bull World Health Organ. 2016 Dec 1;94(12):893-902. doi: 10.2471/BLT.16.173401. Epub 2016 Oct 11. PMID 27994282
- [Background] King C, Boyd N, Walker I, Zadutsa B, Baqui AH, Ahmed S, Islam M, Kainja E, Nambiar B, Wilson I, McCollum ED. Opportunities and barriers in paediatric pulse oximetry for pneumonia in low-resource clinical settings: a qualitative evaluation from Malawi and Bangladesh. BMJ Open. 2018 Jan 30;8(1):e019177. doi: 10.1136/bmjopen-2017-019177. PMID 29382679
- [Background] Emdin CA, Mir F, Sultana S, Kazi AM, Zaidi AK, Dimitris MC, Roth DE. Utility and feasibility of integrating pulse oximetry into the routine assessment of young infants at primary care clinics in Karachi, Pakistan: a cross-sectional study. BMC Pediatr. 2015 Sep 30;15:141. doi: 10.1186/s12887-015-0463-z. PMID 26424473
- [Background] Ginsburg AS, Izadnegahdar R, Klugman KP. World Pneumonia Day 2016: pulse oximetry and oxygen. Lancet Glob Health. 2016 Dec;4(12):e893-e894. doi: 10.1016/S2214-109X(16)30296-0. Epub 2016 Nov 10. No abstract available. PMID 27838358
- [Background] Ginsburg AS, Van Cleve WC, Thompson MI, English M. Oxygen and pulse oximetry in childhood pneumonia: a survey of healthcare providers in resource-limited settings. J Trop Pediatr. 2012 Oct;58(5):389-93. doi: 10.1093/tropej/fmr103. Epub 2011 Dec 14. PMID 22170511
- [Background] Resnicow K, Baranowski T, Ahluwalia JS, Braithwaite RL. Cultural sensitivity in public health: defined and demystified. Ethn Dis. 1999 Winter;9(1):10-21. PMID 10355471
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Baqui AH, Saha SK, Ahmed AS, Shahidullah M, Quasem I, Roth DE, Samsuzzaman AK, Ahmed W, Tabib SM, Mitra DK, Begum N, Islam M, Mahmud A, Rahman MH, Moin MI, Mullany LC, Cousens S, El Arifeen S, Wall S, Brandes N, Santosham M, Black RE; Projahnmo Study Group in Bangladesh. Safety and efficacy of alternative antibiotic regimens compared with 7 day injectable procaine benzylpenicillin and gentamicin for outpatient treatment of neonates and young infants with clinical signs of severe infection when referral is not possible: a randomised, open-label, equivalence trial. Lancet Glob Health. 2015 May;3(5):e279-87. doi: 10.1016/S2214-109X(14)70347-X. Epub 2015 Apr 1. PMID 25841891
- [Background] AFRIcan NEonatal Sepsis Trial Group. Treatment of fast breathing in neonates and young infants with oral amoxicillin compared with penicillin-gentamicin combination: study protocol for a randomized, open-label equivalence trial. Pediatr Infect Dis J. 2013 Sep;32 Suppl 1(Suppl 1 Innovative Treatment Regimens for Severe Infections in Young Infants):S33-8. doi: 10.1097/INF.0b013e31829ff7eb. PMID 23945574
- [Background] Baqui AH, Saha SK, Ahmed AS, Shahidullah M, Quasem I, Roth DE, Williams EK, Mitra D, Shamsuzzaman AK, Ahmed W, Mullany LC, Cousens S, Wall S, Brandes N, Black RE. Safety and efficacy of simplified antibiotic regimens for outpatient treatment of serious infection in neonates and young infants 0-59 days of age in Bangladesh: design of a randomized controlled trial. Pediatr Infect Dis J. 2013 Sep;32 Suppl 1(Suppl 1 Innovative Treatment Regimens for Severe Infections in Young Infants):S12-8. doi: 10.1097/INF.0b013e31829ff790. PMID 23945570
- See also: World Health Organization. Integrated Management of Childhood Illness; Chart Booklet: WHO Library Cataloguin; 2014. — http://apps.who.int/iris/bitstream/handle/10665/104772/9789241506823_Chartbook_eng.pdf;jsessionid=45058111AE386D954C19C57B8AD47E13?sequence=16
- See also: Hauri AM, Armstrong GL, HUTiN YJ. Contaminated injections in health care settings. Comparative quantification of health risks: global and regional burden of disease attributable to selected major risk factors Geneva: World Health Organization. 2003. — http://citeseerx.ist.psu.edu/viewdoc/download?doi=10.1.1.948.7409&rep=rep1&type=pdf#page=1827
- See also: World Health Organization. Revised WHO classification and treatment of pneumonia in children at health facilities: evidence summaries. 2014. — https://www.ncbi.nlm.nih.gov/books/NBK264164/
- See also: Recommendations for management of common childhood conditions: evidence for technical update of pocket book recommendations — http://apps.who.int/iris/bitstream/handle/10665/44774/?sequence=1
- See also: Rall G. Use of a pulse oxymetry sensor device. Google Patents; 1999. — https://patents.google.com/patent/US5911690A/en
- See also: Macefield R. Usability studies and the Hawthorne Effect. Journal of Usability Studies. 2007;2(3):145-54. — http://uxpajournal.org/usability-studies-and-the-hawthorne-effect/
- See also: Smith ID, Coombs SJ. The Hawthorne Effect: is it a help or a hindrance in social science research? Change (Sydney, NSW). 2003;6(1):97. — http://researchspace.bathspa.ac.uk/91/